CLINICAL TRIAL: NCT02893280
Title: Improving Care for Patients With Acute Coronary Syndrome: Acute Coronary Syndrome Sri Lanka Audit Project (ACSSLAP)
Brief Title: Acute Coronary Syndrome Sri Lanka Audit Project
Acronym: ACSSLAP
Status: Withdrawn | Type: Observational
Why Stopped: Due to an incompatibility with the local procedures
Sponsor: University of Colombo (Other)
Collaborators: Ministry of Health, Sri Lanka (Other Government)
Responsible Party: Principal Investigator, Vipula R Bataduwaarachchi, Lecturer in Pharmacology and Pharmacy, University of Colombo
Other Study IDs: UC00101
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Acute Coronary Syndrome; Unstable Angina; Non ST Elevation Myocardial Infarction; ST Elevation Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Aspirin; Clopidogrel; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Enoxaparin; Streptokinase; Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aspirin, clopidogrel, statin, enoxaparin, streptokinase — Acute coronary syndrome treatment
  Other Names: Alteplase

SUMMARY:
ACSSLAP is the first island wide audit project in Sri Lanka on ACS.

DETAILED DESCRIPTION:
Acute coronary syndrome is a leading cause of morbidity and mortality in the world. Even though up-to-date epidemiological data are not available, as per the institutional level experiences this is not differ much in the local settings. Having a free health care system, government of Sri Lanka has to allocate billions of funds and resources from the annual budget for the maintenance of health care system. Being a developing nation this is a considerable burden to the economy of the country. However, prioritization during resource allocation will prevent mal-distribution of limited resources.

Health care system in Sri Lanka should deliver free as well as quality care to the nation. However, lack of updated guidelines in Sri Lanka for the management for acute coronary syndrome (ACS) is a drawback. American College of Cardiology (ACC) and the European Heart Association (EHA) have developed evidence based and most up to date guidelines to standardize clinical practices in the management of ACS. It is recommended to adhere to local or International guidelines to deliver optimal and quality care to ACS patients.

In Sri Lanka, no audits have been conducted in the health sector in relation to patient management practices in the past. Even though institutional level audits have been carried out time to time for the purpose of allocating medicines and other diagnostic resources, island wide large scale audits have not been carried out. Therefore, conducting an audit on health recourse allocation and patient management clinical practices has become a high priority.

Investigators selected ACS as the most important clinical discipline to conduct an audit based on the institutional level data. This audit is included as a well-designed set of clinical criteria derived from the Myocardial Ischemia National Audit Project (MINAP) in UK, SNAPSHOT ACS study in Australia and New Zealand, American College of Cardiology and European Health Association guidelines. These criteria have been extensively reviewed by a panel of cardiologists and physicians to customize it according to the local requirements.

This project will be Coordinated by the Department of Pharmacology, Faculty of Medicine, University of Colombo in collaboration with the Sri Lanka Heart Association, Ceylon College of Physicians and will be carried out through the Quality and safety Unit of the Ministry of Health, Sri Lanka. Funding is sought from the Ministry of Health

ELIGIBILITY:
Inclusion Criteria:

-Patients who are diagnosed with acute coronary syndrome before/after admission to the hospital.

Exclusion Criteria:

* Patient who refuse to give consent
* Patients who are less than 18 years of age
* Patients whose diagnosis later changed to another diagnosis
* Patient who are enrolled in any other study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This audit will be conducted representing the hierarchy of health care delivery system representing tertiary units, teaching hospitals, district general hospitals up to base hospital level where at least a physician is available. Sample size will be considered based on the number of admissions to each hospital. Minimum number from each hospital will be 30. This number was selected as according to International Network on Rational Use of Drugs (INRUD) guidelines of the World Health Organization, a minimum of 30 prescriptions are recommended from each unit and a minimum of 20 units when auditing prescription data to give a minimum of 600 prescription encounters.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Discharge, recovery or death after diagnosed acute coronary syndrome | From the diagnosis of acute coronary syndrome up to 4 weeks of the hospital stay
  Recovery, discharge or death after acute coronary syndrome management following admission to a hospital

OTHER OUTCOMES:
Patient management | From the diagnosis of acute coronary syndrome up to 4 weeks of the hospital stay
  To assess acute coronary sysndrome (ACS) patient management clinical practices island wide
Health care resources utilization | From the diagnosis of acute coronary syndrome up to 4 weeks of the hospital stay
  To assess health care resources utilization for acute coronary syndrome patients island wide

CONTACTS AND LOCATIONS:
Overall Officials: Priyadarshani Galappatthy, MD, Principal Investigator — Department of Pharmacology, Faculty of Medicine, University of Colombo
Locations (1):
- Faculty of Medicine, Colombo, Western Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: Yes
Data will be documented on September 17th, 2016

REFERENCES:
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ; ACC/AHA Task Force Members. 2014 AHA/ACC guideline for the management of patients with non-ST-elevation acute coronary syndromes: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Dec 23;130(25):e344-426. doi: 10.1161/CIR.0000000000000134. Epub 2014 Sep 23. No abstract available. PMID 25249585